CLINICAL TRIAL: NCT01320241
Title: An Unicentric RCT About Novel Radiation Stent Versus Nitinol SEMS for Palliative Treatment of Malignant Biliary Stricture
Brief Title: Radiation Stent Versus Self-expanding Metallic Stents (SEMS) for Palliative Treatment of Malignant Biliary Stricture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Gao-Jun Teng, Director of Department of Radiology, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 320924197612177170-BS
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2011-03

CONDITIONS: Cholangiocellular Carcinoma; Pancreatic Cancer; Gallbladder Cancer; Metastatic Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Gallbladder Neoplasms; Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- novel radiation stent (Active Comparator): Patients undergo placement of a novel biliary stent loaded with 125I seeds on day 1.
  Intervention: Device: self-expandable 125I radioactive seeds-loaded-stent
  Interventions: Device: self-expandable 125I radioactive seeds-loaded-stent
- conventional stent (Experimental): Patients undergo placement of a conventional nitinol SEMS on day1.
  Intervention: Device: self-expandable biliary nitinol alloys stent
  Interventions: Device: self-expandable biliary nitinol alloys stent

INTERVENTIONS:
Device: self-expandable 125I radioactive seeds-loaded-stent — Patients undergo placement of a self-expandable 125I radioactive seeds-loaded-stent on day 1.
  Other Names: irradiation biliary stent
  Arms: novel radiation stent
Device: self-expandable biliary nitinol alloys stent — Patients undergo placement of a conventional self-expandable biliary nitinol alloys stent on day 1.
  Other Names: conventional SEMS
  Arms: conventional stent

SUMMARY:
Malignant biliary obstruction is a common clinical condition caused by various malignancies. Currently,biliary stent implantation guided either by fluoroscopy or endoscopy has become the most important methods for relieving malignant biliary obstruction. However, the benefit for the survival of the patients with palliation of the stent treatment is limited because no therapeutic effects on process of the tumor itself by a stent implantation. Encouraged by the success of 125I esophageal stent in esophageal carcinoma, a novel biliary stent loaded with 125I radioactive seeds has been developed in our institute. After ex vivo and in vivo evaluations for the delivery system, the investigators prospectively compare the responses to treatment with this radiation biliary stent, versus the conventional biliary SEMS in patient with malignant biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Biliary obstruction by any malignant process with histologically or cytologically confirmed by biopsy or previous surgical procedures
* Clinical symptoms of biliary obstruction
* Unresectable or refused to be surgically treated biliary obstruction by any malignant process
* Willing and able to comply with the study procedures and provide written informed consent to participate in the study

Exclusion Criteria:

* Suspected benign bile duct stricture
* Strictures that can not be dilated enough to pass the delivery system
* Perforation of any duct within the biliary tree
* Presence metallic biliary stent or bile duct surgery
* Patients for whom PTC procedures are contraindicated
* Patients with active hepatitis or intrahepatic metastases that extensively involves both lobes of the liver
* Noncooperation or no authorization and signature

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Overall Mean Survival and Median Survival | follow-up in interval of stent insertion and death (3 years)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Technical Success, Clinical Success, Safety (including WBC and Immunological changes of lab, Leakage of the radioactive seeds and Complications related to the procedure. | follow-up in interval of stent insertion and death (3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, MD, PhD, Principal Investigator — Zhong-Da Hospital, Southeast University
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China